CLINICAL TRIAL: NCT01721070
Title: IAP104 - Assessment of Pharmacokinetic Changes Following Concurrent Administration of Sufentanil NanoTab and Ketoconazole in Healthy Subjects
Brief Title: Effect of Ketoconazole on Sufentanil NanoTab Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IAP104
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Pharmacokinetics
Keywords: Area under curve, time to maximum concentration
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUF NT 15 mcg (Experimental): Period 1: One dose of SUF NT 15 mcg administered sublingually. Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
  Interventions: Drug: Sufentanil NanoTab (SUF NT) 15 mcg
- Ketoconazole 400 mg, SUF NT 15 mcg (Experimental): Ketoconazole 400 mg administered once daily for three days. One dose of SUF NT 15 mcg was co-administered sublingually with the third (last) ketoconazole dose.
  Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
  Interventions: Drug: Ketoconazole 400 mg, sufentanil NanoTab (SUF NT) 15 mcg

INTERVENTIONS:
Drug: Sufentanil NanoTab (SUF NT) 15 mcg — Period 1: One dose of SUF NT 15 mcg administered sublingually
  Other Names: SUF NT 15 mcg
  Arms: SUF NT 15 mcg
Drug: Ketoconazole 400 mg, sufentanil NanoTab (SUF NT) 15 mcg — Period 2: Ketoconazole 400 mg administered daily for three days, SUF NT 15 mcg co-administered sublingually on the third day
  Other Names: SUF NT 15 mcg
  Arms: Ketoconazole 400 mg, SUF NT 15 mcg

SUMMARY:
Evaluate the effect of taking ketoconazole on sufentanil plasma concentrations following sublingual administration of sufentanil NanoTab.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking
* Ages 18 to 45 year, inclusive
* BMI between 18 and 30

Exclusion Criteria:

* subjects taking any prescription or OTC medications or vitamins or supplements
* pregnant females
* subjects with pulmonary disease or sleep apnea

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela P. Palmer, MD, PhD, Study Director — Talphera, Inc
Locations (1):
- PRA, Lenexa, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SUF NT 15 mcg Followed by Ketoconazole 400 mg + SUF NT 15 mcg: Period 1: One SUF NT 15 mcg administered sublingually followed by Period 2.
  Period 2: Ketoconazole 400 mg given daily for three days; One SUF NT 15 mcg was also co-administered sublingually with the third (last) ketoconazole dose.
  Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT 15 mcg dosing to block the opioid effects of the sufentanil.
Period: SUF NT 15 mcg
Arm/Group | SUF NT 15 mcg Followed by Ketoconazole 400 mg + SUF NT 15 mcg
Started | 19
Completed | 19
Not Completed | 0
Period: Ketoconazole 400 mg and SUF NT 15 mcg
Arm/Group | SUF NT 15 mcg Followed by Ketoconazole 400 mg + SUF NT 15 mcg
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- SUF NT 15 mcg Then 3 Days of Ketoconazole and SUF NT 15 mcg: Period 1: SUF NT 15 mcg administered once sublingually. Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
  Period 2: Ketoconazole 400 mg given daily for three days. One SUF NT 15 mcg was also co-administered sublingually with the third (last) ketoconazole dose.
  Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
Arm/Group | SUF NT 15 mcg Then 3 Days of Ketoconazole and SUF NT 15 mcg
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants] — Subjects must have been between 18 and 45 years of age, inclusive
  Participants
    <=18 years | 0
    Between 18 and 65 years | 19
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-inf)
Description: Total amount of sufentanil absorbed; After each dosing of Sufentanil NanoTab, serial blood samples will be taken at regular time points.
Time Frame: 0 (pre-dose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 120, 180, 240, 360, 480, 600, 720, and 840 minutes, and 24 hours after dosing.24 hours
Population: 2 of the 19 subjects had incomplete PK data and were excluded from PK analysis (1 due to early withdrawal and 1 due to AE)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- SUF NT 15 mcg: One SUF NT 15 mcg administered sublingually. Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
- Ketoconazole 400 mg and SUF NT 15 mcg: Ketoconazole 400 mg given orally daily for three days. One SUF NT 15 mcg is also co-administered sublingually with the third (last) ketoconazole dose.
  Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
Arm/Group | SUF NT 15 mcg | Ketoconazole 400 mg and SUF NT 15 mcg
Number analyzed (Participants) | 17 | 17
h*pg/mL | 126.47 (46.42) | 223.63 (45.45)

2. Primary Outcome: Cmax
Description: Maximum plasma concentration; After each dosing of Sufentanil NanoTab, serial blood samples will be taken at regular time points.
Time Frame: 0 (pre-dose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 120, 180, 240, 360, 480, 600, 720, and 840 minutes, and 24 hours after dosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Ketoconazole 400 mg and SUF NT 15 mcg: Ketoconazole 400 mg given daily for three days. One SUF NT15 mcg is also co-administered sublingually with the third (last) ketoconazole dose.
  Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
Arm/Group | SUF NT 15 mcg | Ketoconazole 400 mg and SUF NT 15 mcg
Number analyzed (Participants) | 17 | 17
pg/mL | 39.95 (18.57) | 46.00 (16.50)

ADVERSE EVENTS:
Time Frame: Four days
Groups:
- Ketoconazole 400 mg + SUF NT 15 mcg: Ketoconazole 400 mg given daily for three days. One SUF NT 15 mcg was also co-administered sublingually with the third (last) ketoconazole dose.
  Subjects also received one dose of oral naltrexone 50 mg in the evening before and the morning of each SUF NT dosing to block the opioid effects of the sufentanil.
Arm/Group | SUF NT 15 mcg | Ketoconazole 400 mg + SUF NT 15 mcg
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 5/19 | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SUF NT 15 mcg (N=19) | Ketoconazole 400 mg + SUF NT 15 mcg (N=18)
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0
Hot Flush (Vascular disorders) | 1 | 1
Photophobia (Eye disorders) | 0 | 1 — All adverse events listed on this table are included regardless of relationship to study drug (s)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Requires prior approval from AcelRx Pharmaceuticals, Inc.